CLINICAL TRIAL: NCT02110875
Title: Strength and Balance in Gender- and Age-Matched Controls: SubStudy to "The Effects of Vitamin D on Balance in Parkinson's Disease"
Brief Title: Strength and Balance in Gender- and Age-Matched Controls
Acronym: VITDC
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amie Peterson, MD, Assistant Professor, Oregon Health and Science University
Other Study IDs: e9576
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CONTROLS: Age- and Gender-Matched Controls

SUMMARY:
The purpose of this study is to learn more about balance and strength in an elderly population (60 and older). Data will be compared between controls and the age/gender- matched PD participants in study "The Effects of vitamin D on Balance in Parkinson's disease" (OHSU IRB # 6482). Specifically a t-test will be used to compare total work and total power on leg extension and flexion, composite SOT score conditions 1-3 and 4-6, response strength and latency on MCT, and turn duration from the iMOBILITY between the two groups.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Over the age of 59
* Gender and Age-Matched (within 3 years) of main protocol participants

Exclusion Criteria:

* Parkinson's disease diagnosis
* Significant cognitive deficits.
* Another neurological or orthopedic deficit that in the investigator's opinion would have a significant impact on gait and cognition (e.g. stroke, fracture).

This study involves one visit to Oregon Health & Science University. The study visit will last approximately 2 hours.

Measurements:

1. The participant's balance will be assessed by having them stand on a platform and completing mental tasks such as naming the alphabet backwards. They will be asked to have their eyes open on some tasks and closed on other tasks. For safety, they will wear a harness like those used by rock climbers.
2. The participant's ability to move and balance will be measured by putting six sensors on their bodies (both wrists, both ankles, chest, and back). Each sensor is about the size and weight of a deck of cards. To measure movement and balance, participants will rise from a chair, walk three feet, turn around, walk back to the chair, and sit down.
3. The participant's strength will be evaluated using a machine that resembles a stationary exercise bike. They will have one leg and foot strapped onto the machine. Participants will then be asked to flex and extend their leg as quickly as possible five times. This will be repeated with the other leg.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 59
* Gender and Age-Matched (within 3 years) of main protocol participants

Exclusion Criteria:

* Parkinson's disease diagnosis
* Significant cognitive deficits.
* Another neurological or orthopedic deficit that in the investigator's opinion would have a significant impact on gait and cognition (e.g. stroke, fracture).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Elderly (over 59 years old) without Parkinson's disease or Parkinsonism.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Strength (BIODEX) | Visit 1
  The participant's strength will be evaluated using a machine that resembles a stationary exercise bike. They will have one leg and foot strapped onto the machine. Participants will then be asked to flex and extend their leg as quickly as possible five times. This will be repeated with the other leg.

SECONDARY OUTCOMES:
Balance (SOT) | Visit 1
  The participant's balance will be assessed by having them stand on a platform and completing mental tasks such as naming the alphabet backwards. They will be asked to have their eyes open on some tasks and closed on other tasks. For safety, they will wear a harness like those used by rock climbers.

CONTACTS AND LOCATIONS:
Overall Officials: Amie L Peterson, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Moreland JD, Richardson JA, Goldsmith CH, Clase CM. Muscle weakness and falls in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2004 Jul;52(7):1121-9. doi: 10.1111/j.1532-5415.2004.52310.x. PMID 15209650
- [Background] Horlings CG, van Engelen BG, Allum JH, Bloem BR. A weak balance: the contribution of muscle weakness to postural instability and falls. Nat Clin Pract Neurol. 2008 Sep;4(9):504-15. doi: 10.1038/ncpneuro0886. PMID 18711425
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Inkster LM, Eng JJ, MacIntyre DL, Stoessl AJ. Leg muscle strength is reduced in Parkinson's disease and relates to the ability to rise from a chair. Mov Disord. 2003 Feb;18(2):157-62. doi: 10.1002/mds.10299. PMID 12539208
- [Background] Allen NE, Canning CG, Sherrington C, Fung VS. Bradykinesia, muscle weakness and reduced muscle power in Parkinson's disease. Mov Disord. 2009 Jul 15;24(9):1344-51. doi: 10.1002/mds.22609. PMID 19425085